CLINICAL TRIAL: NCT01178411
Title: An Extension Protocol for Subjects Who Were Previously Enrolled in Other Tivantinib (ARQ 197) Protocols
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-299; 2010-020151-31 (EudraCT Number)
Record Dates: First submitted 2010-07-21; First posted 2010-08-10 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Advanced Solid Tumors
Keywords: hepatocellular carcinoma; renal cell carcinoma; melanoma; non-small cell lung cancer; breast cancer; ovarian cancer; MiT tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Melanoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Ovarian Neoplasms | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tivantinib (Monotherapy or Combination Therapy) (Experimental): Tivantinib 360 mg will be administered twice daily, orally, with meals, as a monotherapy or in combination with other drug therapies.
  Interventions: Drug: Tivantinib; Drug: Anti-Cancer Combination Therapy

INTERVENTIONS:
Drug: Tivantinib — Tivantinib 360 mg (3 x 120 mg tablets or capsules) twice daily by mouth.
  Other Names: ARQ 197
Drug: Anti-Cancer Combination Therapy — Tivantinib 360 mg twice daily in combination with other anti-cancer therapy (eg, erlotinib,sorafenib, pemetrexed, docataxel, gemcitabine, irinotecan, and/or cetuximab) at the same dose and schedule in which they were administered in the original (previous) study.
  Other Names: ARQ 197

SUMMARY:
This is an extension study that will allow participants to continue to receive study therapy when the original studies into which they were enrolled have reached their designated end-dates. This extension study is designed to further evaluate the safety and tolerability of tivantinib (ARQ 197) monotherapy or in combination with other drug(s) when given to participants who tolerated previous treatment well and may benefit from the continuing treatment.

DETAILED DESCRIPTION:
This open label extension protocol enrolls participants who were treated in previous phase 1 (NCT01149720, NCT01517399, NCT01699061, NCT00612703, NCT00827177, and NCT00874042) and phase 2 (NCT00777309, NCT00557609, NCT00988741, NCT01395758 , and NCT01055067) tivantinib studies that have reached their designated end-dates. Participants enrolled in this extension protocol will provide further safety and tolerability information about tivantinib monotherapy or in combination with other drug(s) at the same dose(s), and same schedule(s) in which they were originally enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent to participate in clinical study of tivantinib
* Male or female participants of the age defined in the original protocol they were enrolled.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤3 (or ≤2 for tivantinib-naive participants)
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
  * Hemoglobin ≥8.0 g/dL (or ≥ 9.0 g/dL for tivantinib-naïve participants)
* Enrollment within 14 days of the completion of End of Treatment Visit of the original study
* Participants, who participated in previous ARQ 197 studies that have reached their designated end-dates, who did not meet discontinuation criteria in their original study, and who may, in the opinion of the Investigator and the Sponsor, benefit from treatment
* Women of childbearing potential must have a negative pregnancy test performed within 14 days of the start of study drug. Both men and women enrolled in this study must agree to use adequate birth control measures while on study

Exclusion Criteria:

* Known or suspected allergy to ARQ 197
* Substance abuse, medical, psychological or social conditions that may interfere with the participant's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the participant and his/her compliance in the study
* A serious uncontrolled medical disorder/condition that in the opinion of the Investigator would impair the ability of the participant to receive protocol therapy
* Requirement to receive other concurrent chemotherapy (excluding combination therapy defined in original protocol), immunotherapy, radiotherapy, or any other investigational drug while on study. Palliative radiotherapy is allowed provided that:

  * in the opinion of the Investigator, the participant does not have progressive disease
  * the radiation field does not encompass a target lesion
  * no more than 10% of the participant's bone marrow is irradiated

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08-31 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants previously enrolled in phase 1 or phase 2 studies of tivantinib (ARQ 197) were eligible for enrollment.
Groups:
- Tivantinib (Monotherapy or Combination): Participants received tivantinib 360 mg twice daily by mouth as monotherapy or combination therapy.
Period: Overall Study
Arm/Group | Tivantinib (Monotherapy or Combination)
Started | 60
Completed | 0
Not Completed | 60
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 1
Not completed — Progressive disease per RECIST | 32
Not completed — Progressive disease per clinician | 9
Not completed — Physician Decision | 6
Not completed — Death | 1
Not completed — No reason provided | 1
Not completed — Drug manufacturing ended | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tivantinib (Monotherapy or Combination)
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (14.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 54
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Extent of Exposure to ARQ 197 in Participants Benefiting From Prior ARQ 197 Therapy
Description: The duration of ARQ 197 exposure in this study was calculated as [(date of last dose of study drug - date of first dose of study drug) + 1]. Results refer to duration of ARQ 197 treatment in the present study only (i.e., does not include treatment received during participation in "feeder" studies).
Time Frame: Up to 3,021 days (up to 14-Jan-2019)
Population: All participants who received ≥1 dose of study drug are included.
Measure: Median (Full Range); unit: Days
Arm/Group | Tivantinib (Monotherapy or Combination)
Number analyzed (Participants) | 60
Days | 125 [5 to 3021]

2. Secondary Outcome: Number of Participants With ≥1 Treatment-emergent Adverse Event (TEAE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 3021 days
Population: All participants who received ≥1 dose of study drug are included.
Measure: Number; unit: Participants
Arm/Group | Tivantinib (Monotherapy or Combination)
Number analyzed (Participants) | 60
Participants | 56

3. Secondary Outcome: Number of Participants Discontinuing Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to 3,021 days
Population: All participants who received ≥1 dose of study drug are included.
Measure: Number; unit: Participants
Arm/Group | Tivantinib (Monotherapy or Combination)
Number analyzed (Participants) | 60
Participants | 6

ADVERSE EVENTS:
Time Frame: Up to 3021 days
Description: All participants who received ≥1 dose of study drug are included.
Arm/Group | Tivantinib (Monotherapy or Combination)
All-Cause Mortality (participants affected / at risk) | 4/60
Serious Adverse Events (participants affected / at risk) | 19/60
Other Adverse Events (participants affected / at risk) | 55/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivantinib (Monotherapy or Combination) (N=60)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Abdominal mass (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fractured Sacrum (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Radical neck dissection (Surgical and medical procedures) | 1
Thrombectomy (Surgical and medical procedures) | 1
Aortic stenosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Superior vena caval occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tivantinib (Monotherapy or Combination) (N=60)
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 20
Fatigue (General disorders) | 17
Mucosal inflammation (General disorders) | 5
Oedema peripheral (General disorders) | 7
Pain (General disorders) | 7
Pyrexia (General disorders) | 5
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 7
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 6
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall have the right to publish the results of research performed under this protocol, provided that such publication does not disclose any confidential information or trade secrets of ArQule (other than the data).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT01178411/Prot_SAP_000.pdf